CLINICAL TRIAL: NCT03701984
Title: The Effect of Intrauterine Lidocaine Infusion and Oral Tramadol on Pain During Diagnostic Office Hysteroscopy in Postmenopausal Women: Randomized Double-Blind Controlled Study
Brief Title: The Effect of Intrauterine Lidocaine Infusion and Oral Tramadol on Pain During Diagnostic Office Hysteroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: hysteroscopy
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — Lidocaine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lidocaine infusion arm (Experimental): The lidocaine group will be administered a 1,000 ml distention medium containing 5 ml lidocaine per 250 ml (DEBOCAINE (LIDOCAINE) 2% 1 VIAL 50 ML, Sigma-Tec pharmaceutical Industry. Co. Egypt) and oral placebo similar to tramadol(given 1 hour before the procedure).
  Interventions: Drug: Lidocaine
- tramadol arm (Active Comparator): will be administered with an oral tramadol tablet (Tramal®, Memphis, Giza, Egypt) 1 h before the procedure and with a 1,000 ml distention medium containing 5 ml serum physiologic per 250 ml.
  Interventions: Drug: Tramadol
- placebo group (Placebo Comparator): will be administered with a 1,000 ml distention medium containing 5 ml serum physiologic per 250 ml and oral placebo(1 h before the procedure).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lidocaine — The lidocaine group will be administered a 1,000 ml distention medium containing 5 ml lidocaine per 250 ml (DEBOCAINE (LIDOCAINE) 2% 1 VIAL 50 ML, Sigma-Tec pharmaceutical Industry. Co. Egypt) and oral placebo similar to tramadol(given 1 hour before the procedure).
  Other Names: lidocaine infusion arm
  Arms: lidocaine infusion arm
Drug: Tramadol — an oral tramadol tablet (Tramal®, Memphis, Giza, Egypt) 1 h before the procedure and with a 1,000 ml distention medium containing 5 ml serum physiologic per 250 ml.
  Other Names: tramadol HCL arm
  Arms: tramadol arm
Drug: placebo — a 1,000 ml distention medium containing 5 ml serum physiologic per 250 ml and oral placebo(1 h before the procedure).
  Other Names: placebo arm
  Arms: placebo group

SUMMARY:
The purpose of this study is to compare the effectiveness of Tramadol and intrauterine lidocaine infusion in reducing pain during outpatient diagnostic hysteroscopy in postmenopausal women.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of Tramadol and intrauterine lidocaine infusion in reducing pain during outpatient diagnostic hysteroscopy in postmenopausal women. Postmenopausal Women undergoing outpatient hysteroscopy in Cairo university will be divided into three groups, the first group will receive Tramadol 5mg 1 hour before the procedure, the second group will receive 20 ml lidocaine in 1000 ml normal saline infusion during the procedure, and the third will receive a placebo. A visual analog scale will assess pain.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal patients with an indication for office hysteroscopy (postmenopausal bleeding or abnormal ultrasound findings)
* Consent to the procedure

Exclusion Criteria:

* Positive Chlamydia culture.
* patients who have an Allergy to local anesthesia or tramadol.
* A previous adverse reaction to any of the drugs used in the study.
* Patients were receiving any form of analgesia or current use of monoamine oxidase inhibitors.
* Nulliparous patients and patients with cervical pathology, retroverted uterus (detected by transvaginal ultrasound), and previous cervical surgery.
* Patients who have severe vaginal bleeding.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Pain perception during the procedure | 10 minutes after starting the procedure.
  The pain will be assessed using a visual analogue scale(VAS) after inserting the hysteroscope through the cervical canal.VAS of 0 indicates no pain and VAS of 10 indicates the worst possible experienced pain. The pain VAS is self-completed by the patients. The patients are asked to place a line perpendicular to the VAS line at the point that represents their pain intensity

SECONDARY OUTCOMES:
Pain perception after the procedure | 10 minutes after the procedure.
  Pain will be assessed using a visual analog scale(VAS) 10 minutes after the procedure.
  VAS of 0 indicates no pain and VAS of 10 indicates the worst possible experienced pain.
  The pain VAS is self-completed by the patient. The patients are asked to place a line perpendicular to the VAS line at the point that represents their pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: AHMED S ASHOUR, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine Cairo university, Giza, Egypt

REFERENCES:
- [Derived] Samy A, Nabil H, Abdelhakim AM, Mahy ME, Abdel-Latif AA, Metwally AA. Pain management during diagnostic office hysteroscopy in postmenopausal women: a randomized study. Climacteric. 2020 Aug;23(4):397-403. doi: 10.1080/13697137.2020.1742685. Epub 2020 Apr 17. PMID 32299254